CLINICAL TRIAL: NCT04622995
Title: Exploring the Utility and Safety of Benzodiazepine Prescribing Among People Receiving Opiate Replacement Therapy in Scotland (the BENZORT Study).
Brief Title: Benzodiazepines in Opiate Replacement Therapy
Acronym: BENZORT
Status: Completed | Type: Observational
Sponsor: University of Stirling (Other)
Collaborators: NHS Research Scotland (Other)
Responsible Party: Principal Investigator, Joe Schofield, Research Fellow, University of Stirling
Other Study IDs: BENZORT
Record Dates: First submitted 2020-11-03; First posted 2020-11-10 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Substance-Related Disorders
Keywords: Benzodiazepine; Opiate Replacement Treatment; Drug-Related Death; Overdose
MeSH Terms: conditions — Substance-Related Disorders; Drug Overdose | interventions — Benzodiazepines; Diazepam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed: Patients prescribed opiate replacement therapy plus a benzodiazepine.
  Interventions: Drug: Benzodiazepine
- Unexposed: Patients prescribed opiate replacement therapy with no benzodiazepine prescribing.

INTERVENTIONS:
Drug: Benzodiazepine — Benzodiazepine prescribing
  Other Names: Valium; Diazepam
  Groups: Exposed

SUMMARY:
Drug-related deaths (DRD) are a significant and increasing public health problem in Scotland. Benzodiazepines and BZD-type substances (BZD) are increasingly implicated in DRD. In 2018, BZDs were implicated in 67% of DRD, often in combination with other illicit and prescribable substances including Opiate Replacement Therapies (ORT) such as methadone and buprenorphine.

Illicit BZD use and dependence is higher among people with other substance use disorders. 29% of patients presenting to Scottish addiction services report current illicit BZD use. There is widespread variance in approaches to the clinical management of BZD dependence among people with opioid use disorder in Scotland. Some addiction clinicians are reluctant to prescribe BZD to people on ORT, some will prescribe BZD with the primary aim of dose reduction and detoxification, others will consider longer-term maintenance prescribing whilst patients stabilise on ORT.

Previous research has identified increased risks of mortality among people taking BZD and ORT. Other work suggests that co-prescribing BZD and ORT increases patient engagement and retention in addiction treatment.

This retrospective cohort study will analyse anonymised, linked data on people who received ORT between 01/01/2010 and 31/12/2020 to explore any relationships between exposure (co-prescribing of BZD and ORT) and harms including: mortality (all-cause and DRD), hospitalisation, illicit drug use during ORT, and reduced retention in addiction care.

DETAILED DESCRIPTION:
Scotland is experiencing a 'public health emergency' of escalating drug-related deaths (DRD) in which benzodiazepine (BZD) are increasingly implicated, often in combination with other substances (National Records of Scotland, 2019; Scottish Government, 2019).

In 2008 BZD were implicated in 26% (n=149) of DRD and were exclusively prescribable drugs such as diazepam, although the source is not known. By 2018 BZD and BZD-type drugs were implicated in 67% (792) of DRD, predominately substances not available on prescription in the United Kingdom (UK) such as etizolam and alprazolam (Xanax). We refer to these as illicit BZD.

People who use illicit BZD, of unknown constituents and potency, can inadvertently or deliberately consume megadoses of BZD many times in excess of safe therapeutic doses, often with alcohol and other drugs, which combine to increase the risk of harm and death. Rights, Respect and Recovery, the current drug and alcohol strategy, expressed Scottish Government concern regarding the increased prevalence and potency of BZD-type drugs.

People presenting to addiction services for initial assessment frequently report illicit BZD use in the month prior to assessment, an average of 2,561 (29%) per year in the past five years for which data are available. The prevalence of illicit BZD use is known to be higher among people with other substance use disorders, especially problematic opiate and/or alcohol dependence. A systematic review identified a high prevalence (typically >40%) among people on Opiate Replacement Therapy (ORT).

The picture of BZD prescribing among people on ORT is complex and evolving. Previous work shows that BZD prescribing among ORT patients is associated with increased harms including mortality, but conversely protective factors such as increased engagement in care. Scottish addiction specialists have confirmed that some addiction services are exploring maintenance prescribing to reduce the risks associated with illicit BZD use among ORT patients. However clinical guidance does not currently provide a framework for this. Evidence of patient safety and other outcomes from BZD prescribing in the context of ORT is sparse and conflicting. A 2018 Cochrane review concluded "it is not possible to draw firm conclusions regarding pharmacological interventions to facilitate BZD discontinuation in chronic BZD users". Recent UK public health alerts have highlighted the need for caution and additional monitoring when co-prescribing BZD and ORT, and the need for improved harm reduction advice regarding the risk of illicit BZD. Addiction clinicians have indicated there has been disagreement among certifying pathologists regarding the role of benzodiazepines in DRD.

There is a need to understand patterns of, and outcomes from, BZD prescribing among ORT patients in Scotland to inform safe and effective clinical practice, address problematic BZD use in the content of poly-drug use, and reduce the risk of harms including mortality among people who use drugs (PWUD).

ELIGIBILITY:
The cohort will consist of people who were prescribed ORT between 01/01/2010 and 31/12/2020. The definition of ORT is based on the following medications and associated British National Formulary (BNF) codes:

Chemical (BNF code): Buprenorphine Hydrochloride/Naloxone Hydrochloride (0410030B0); Buprenorphine Hydrochloride (0410030A0); Methadone Hydrochloride (0410030C0)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population includes people who received medication assisted treatment for the management of opiate / opioid addiction from community settings (e.g. community-based specialist addiction services and primary care physicians 'General Practitioners').
Sampling Method: Non-Probability Sample
Enrollment: 46899 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | From enrollment to end December 2020
  Death from any cause

SECONDARY OUTCOMES:
Drug-related death | From enrollment to end December 2020
  Fatal drug overdose
Drug overdose (non-fatal) | From enrollment to end December 2020
  Non-fatal drug overdose
Hospitalisation | From enrollment to end December 2020
  Admission to hospital from any cause
Evidence of illicit drug use during Opiate Substitution Therapy | From enrollment to end December 2020
  Evidence of illicit drug use during Opiate Substitution Therapy
Retention in care | From enrollment to end December 2020
  Retention in specialist addiction care for substance use disorder(s)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Schofield, MPH, Principal Investigator — University of Stirling
Locations (1):
- NHS Scotland, Edinburgh, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baandrup L, Ebdrup BH, Rasmussen JO, Lindschou J, Gluud C, Glenthoj BY. Pharmacological interventions for benzodiazepine discontinuation in chronic benzodiazepine users. Cochrane Database Syst Rev. 2018 Mar 15;3(3):CD011481. doi: 10.1002/14651858.CD011481.pub2. PMID 29543325
- [Background] Bakker A, Streel E. Benzodiazepine maintenance in opiate substitution treatment: Good or bad? A retrospective primary care case-note review. J Psychopharmacol. 2017 Jan;31(1):62-66. doi: 10.1177/0269881116675508. Epub 2016 Dec 14. PMID 28072037
- [Background] Chen KW, Berger CC, Forde DP, D'Adamo C, Weintraub E, Gandhi D. Benzodiazepine use and misuse among patients in a methadone program. BMC Psychiatry. 2011 May 19;11:90. doi: 10.1186/1471-244X-11-90. PMID 21595945
- [Background] Cornish R, Macleod J, Strang J, Vickerman P, Hickman M. Risk of death during and after opiate substitution treatment in primary care: prospective observational study in UK General Practice Research Database. BMJ. 2010 Oct 26;341:c5475. doi: 10.1136/bmj.c5475. PMID 20978062
- [Background] Macleod J, Steer C, Tilling K, Cornish R, Marsden J, Millar T, Strang J, Hickman M. Prescription of benzodiazepines, z-drugs, and gabapentinoids and mortality risk in people receiving opioid agonist treatment: Observational study based on the UK Clinical Practice Research Datalink and Office for National Statistics death records. PLoS Med. 2019 Nov 26;16(11):e1002965. doi: 10.1371/journal.pmed.1002965. eCollection 2019 Nov. PMID 31770388
- [Background] McCowan C, Kidd B, Fahey T. Factors associated with mortality in Scottish patients receiving methadone in primary care: retrospective cohort study. BMJ. 2009 Jun 16;338:b2225. doi: 10.1136/bmj.b2225. PMID 19535400
- [Background] Park TW, Larochelle MR, Saitz R, Wang N, Bernson D, Walley AY. Associations between prescribed benzodiazepines, overdose death and buprenorphine discontinuation among people receiving buprenorphine. Addiction. 2020 May;115(5):924-932. doi: 10.1111/add.14886. Epub 2020 Jan 20. PMID 31916306
- [Background] Votaw VR, Geyer R, Rieselbach MM, McHugh RK. The epidemiology of benzodiazepine misuse: A systematic review. Drug Alcohol Depend. 2019 Jul 1;200:95-114. doi: 10.1016/j.drugalcdep.2019.02.033. Epub 2019 May 7. PMID 31121495
- [Background] Scottish Government. (2019). Statistics show highest ever level of drug deaths. Scottish Government. Edinburgh. Retrieved from https://news.gov.scot/news/statistics-show-highest-ever-level-of-drug-deaths
- [Background] Scottish Government. (2018). Rights, Respect and Recovery. Edinburgh. Retrieved from https://www.gov.scot/binaries/content/documents/govscot/publications/strategy-plan/2018/11/rights-respect-recovery/documents/00543437-pdf/00543437-pdf/govscot%3Adocument/00543437.pdf
- [Background] Public Health England; (2020, July 24). Evidence of harm from illicit or fake benzodiazepines. Retrieved October 16, 2020, from https://www.cas.mhra.gov.uk/ViewandAcknowledgment/ViewAlert.aspx?AlertID=103075
- [Background] National Records of Scotland. (2019). Drug-related Deaths in Scotland in 2018. Edinburgh: National Records of Scotland. Retrieved from https://www.nrscotland.gov.uk/statistics-and-data/statistics/statistics-by-theme/vital-events/deaths/drug-related-deaths-in-scotland/2018
- [Background] Medicines and Healthcare products Regulatory Agency. (2020, March 18). Benzodiazepines and opioids: reminder of risk of potentially fatal respiratory depression. Retrieved October 16, 2020, from https://www.gov.uk/drug-safety-update/benzodiazepines-and-opioids-reminder-of-risk-of-potentially-fatal-respiratory-depression
- [Background] Johnson, C. F., Barnsdale, L. R., & McAuley, A. (2016). Investigating the role of benzodiazepines in drug-related mortality: a systematic review undertaken on behalf of the Scottish National Forum on Drug-Related Deaths. Retrieved from https://www.scotpho.org.uk/media/1159/scotpho160209-investigating-the-role-of-benzodiazepines-in-drug-related-mortality.pdf
- [Background] Information Services Division. (2020). Scottish Drug Misuse Database: Overview of Initial Assessments for Specialist Drug Treatment 2018/19. Edinburgh. Retrieved from https://beta.isdscotland.org/find-publications-and-data/lifestyle-and-behaviours/substance-use/scottish-drug-misuse-database/3-march-2020/
- [Background] EMCDDA. The misuse of benzodiazepines among high-risk opioid users in Europe, Perspectives on drugs (2018). Portugal. Retrieved from http://www.emcdda.europa.eu/topics/pods/benzodiazepines_en
- [Derived] Best CS, Matheson C, Robertson J, Ritchie T, Cowden F, Dumbrell J, Duncan C, Kessavalou K, Woolston C, Schofield J. Association between benzodiazepine coprescription and mortality in people on opioid replacement therapy: a population-based cohort study. BMJ Open. 2024 Mar 14;14(3):e074668. doi: 10.1136/bmjopen-2023-074668. PMID 38485490